CLINICAL TRIAL: NCT00772915
Title: A Phase II Trial of Revlimid® and "On Demand" Dexamethasone Dosing in Patients With Newly Diagnosed Symptomatic Multiple Myeloma
Brief Title: Lenalidomide With or Without Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000616057; P30CA015083 (NIH); MC0884 (Other: Mayo Clinic Cancer Center); 08-002093 (Other: Mayo Clinic IRB); NCI-2009-01201 (Registry Identifier: NCI CTRP); RV-MM-PI-367 (Other: Celgene Protocol)
Record Dates: First submitted 2008-10-12; First posted 2008-10-15 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide with On-Demand Dexamethasone (Experimental): Lenalidmoide: 25mg once daily orally with food on days 1-21 of 28 day cycle until progression or to a maximum of 18 cycles.
  Dexamethasone: 10-40 mg once weekly (days 1, 8, 15, & 22) orally with food until progression.
  Interventions: Drug: dexamethasone; Drug: lenalidomide

INTERVENTIONS:
Drug: dexamethasone — Dose: -40 mg once weekly (days 1, 8, 15, & 22) orally with food until progression.
  If after 3 cycles, a partial response is not achieved on lenalidomide alone, dexamethasone 10 mg weekly will be added, and the weekly dexamethasone dose will be increased by 10 mg each cycle to a maximum of 40 mg weekly, as long as a partial response is not achieved. If a partial response is achieved at a dose of dexamethasone less than 40 mg weekly, patients will continue on that dose. If progression at any time, increase dexamethasone to 40 mg weekly. Patient will go off study only when progression is documented while receiving 40 mg/week of dexamethasone or the maximum tolerated dose of dexamethasone (if prior dose reductions have been implemented for toxicity). Increases in dexamethasone dose are to be made only at the initiation of a cycle.
  If progression at any time while on lenalidomide alone (first 3 cycles), add dexamethasone 40 mg weekly.
Drug: lenalidomide — 25mg once daily orally with food on days 1-21 of 28 day cycle until progression or to a maximum of 18 cycles.
  Lenalidomide alone will be administered for the first 3 cycles, then in combination with dexamethasone as needed (described).

SUMMARY:
RATIONALE: Lenalidomide and dexamethasone may stop the growth of multiple myeloma by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well lenalidomide works with or without dexamethasone in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the progression-free survival at 1 year in patients with newly diagnosed symptomatic multiple myeloma treated with lenalidomide alone or in combination with dexamethasone added for disease progression or lack or partial response.

Secondary

* To assess the response rate of this regimen in these patients.
* To assess the toxicity of this regimen in these patients.

Tertiary

* To examine the effect of lenalidomide alone on tumor specific immunity and global parameters of immune function.
* To examine the effect of dexamethasone addition in patients requiring steroids.
* To correlate changes in parameters of immune response and measures of disease response.
* To examine the antiangiogenic activity of lenalidomide alone and in combination with dexamethasone.
* To examine the effect of lenalidomide alone on tumor cell survival and proliferation.

OUTLINE: Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for up to 18 courses in the absence of second disease progression or unacceptable toxicity. Beginning in course 4, patients experiencing stable or progressive disease also receive concurrent oral dexamethasone once daily on days 1, 8, 15, and 22 and for all subsequent courses.

Blood and bone marrow samples are collected periodically for pharmacological and correlative studies. Samples are analyzed for parameters of immune activation, cell proliferation and apoptosis, and circulating tumor cells and endothelial cells via flow cytometry; global impact of therapy on immune cell subsets via immunophenotype analysis; and angiogenesis via CD34 staining.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed multiple myeloma, meeting the following criteria:

  * Symptomatic disease
  * Previously untreated disease
* Measurable or evaluable disease, defined by ≥ 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g/dL
  * Monoclonal protein > 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa:lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
  * Measurable soft tissue plasmacytoma, not previously radiated
* No monoclonal gammopathy of unknown significance or asymptomatic myeloma

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 (PS 3 allowed if secondary to pain)
* ANC ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective forms of contraception 28 days prior to, during and 28 days after study treatment
* Registered into the RevAssist® program and willing to comply with program requirements
* Able to take prophylactic aspirin (325 mg/day) or warfarin or low molecular weight heparin
* Willing to provide mandatory blood and bone marrow samples
* Willing to return for follow up
* No uncontrolled infection
* No NYHA class III or IV heart failure
* No active deep vein thrombosis that has not been therapeutically anticoagulated
* No known hypersensitivity to thalidomide
* No known HIV positivity
* No known hepatitis type A, B, or C infection
* No other prior active malignancy within the past 2 years, except currently treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior radiotherapy for solitary plasmacytoma
* More than 28 days since other prior experimental drug or therapy
* Prior clarithromycin, DHEA, anakinra, pamidronate, or zoledronic acid allowed
* No prior lenalidomide
* No prior cytotoxic chemotherapy
* No prior corticosteroids (≥ 160 mg of dexamethasone or equivalent) for this disease

  * Prior corticosteroid for nonmalignant disease allowed
  * Concurrent corticosteroids allowed (≤ 20 mg/day of prednisone or equivalent)
* Concurrent palliative radiotherapy for bone pain or fracture allowed
* No other concurrent anticancer agents or treatments

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-nine (39) participants were recruited at Mayo Clinic (Rochester) between December 2008 and April 2010.
Pre-assignment Details: One participant canceled prior to starting treatment; this participant has been removed from all analyses.
Groups:
- Lenalidomide With On-Demand Dexamethasone: Lenalidomide: 25mg once daily orally with food on days 1-21 of 28 day cycle until progression or to a maximum of 18 cycles.
  Dexamethasone: 10-40 mg once weekly (days 1, 8, 15, & 22) orally with food until progression.
Period: Overall Study
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Started | 38
Completed | 23
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 38
Durie Salmon Stage at Diagnosis [Number; unit: participants]
  Stage I: Low Cell Mass | 8
  Stage II: Intermediate Cell Mass | 15
  Stage III: High Cell Mass | 12
  Not Assessed | 3
Parameter of Hematologic Response: Serum M-Spike >= 1 mg/dL [Number; unit: participants]
  Yes | 26
  No | 12
Parameter of Hematologic Response: Serum Immunoglobulin Free Light Chain >= 10 mg/dL [Number; unit: participants]
  Yes | 25
  No | 13
Parameter of Hematologic Response: Urine M-Spike >= 200 mg/24 hours [Number; unit: participants]
  Yes | 14
  No | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 12 Months
Description: PFS rate at 12 months is defined as the percentage of participants who are alive and progression-free at 12 months. Progression is exclusively defined as a patient with progressive disease while receiving treatment with lenalidomide in combination with dexamethasone. Progression was defined as any one or more of the following: An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
Time Frame: 12 months from registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
percentage of participants | 79 [65 to 96]

2. Secondary Outcome: Confirmed Response Rate
Description: Confirmed response rate is defined as the percentage of participants who achieved a response that was confirmed on 2 consecutive evaluations during treatment
  * Complete Response(CR): Complete disappearance of M-protein from serum & urine on immunofixation, normalization of Free Light Chain (FLC) ratio & <5% plasma cells in bone marrow (BM)
  * Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <100 mg per 24 hours; <=5% plasma cells in BM
  * Partial Response PR): >= 50% reduction in serum M-Component and/or Urine M-Component >= 90% reduction or <200 mg per 24 hours; or >= 50% decrease in difference between involved and uninvolved FLC levels
Time Frame: Up to 18 cycles from registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
percentage of participants | 61 [43 to 76]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from registration to death of any cause. Participants were followed for a maximum of 3 years from randomization. The median OS with 95% CI was estimated using the Kaplan Meier method
Time Frame: Time from registration to death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
months | 61.1 [26 to 75]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from registration to progression or death due to any cause. The median PFS with 95%CI was estimated using the Kaplan Meier method.
  Progression was defined as any one or more of the following:An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
Time Frame: Time from registration to progression or death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
months | 27 [13.7 to 75]

5. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Event at Least Possibly Related to Treatment (Toxicity)
Description: The number of participants who experienced toxicity (defined as at least one grade 3 or higher adverse event at least possibly related to treatment) is reported below.
Time Frame: Duration on treatment (up to 18 cycles from registration)
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Number analyzed (Participants) | 38
Participants | 23

ADVERSE EVENTS:
Groups:
- Lenalidomide With On-Demand Dexamethasone: Dexamethasone: 10-40 mg once weekly (days 1, 8, 15, & 22) orally with food until progression.
Arm/Group | Lenalidomide With On-Demand Dexamethasone
Serious Adverse Events (participants affected / at risk) | 9/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide With On-Demand Dexamethasone (N=38)
Left ventricular failure (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide With On-Demand Dexamethasone (N=38)
Anemia (Blood and lymphatic system disorders) | 36 (311)
Cataract (Eye disorders) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (9)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 34 (258)
Pain (General disorders) | 1 (1)
Pain-Chest (General disorders) | 2 (2)
Gallbladder (cholecystitis) infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Skin (cellulites) infection (Infections and infestations) | 2 (2)
Upper airway infection (Infections and infestations) | 3 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Bilirubin (Investigations) | 2 (4)
Creatinine increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 33 (174)
Lymphocyte count decreased (Investigations) | 3 (12)
Neutrophil count decreased (Investigations) | 31 (171)
Platelet count decreased (Investigations) | 19 (108)
Weight gain (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (150)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (3)
Depression (Psychiatric disorders) | 1 (8)
Insomnia (Psychiatric disorders) | 3 (3)
Renal Failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flashes (Vascular disorders) | 1 (2)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes